CLINICAL TRIAL: NCT01206361
Title: Persistence Of Use Of Topical Prostaglandin Fixed Dose Combination In The United Kingdom Primary Care: An Observational Study In Thin
Brief Title: Real World Data Study Assessing The Persistency Of Xalacom And The Other Fixed Dose Combination Products, Duotrav And Ganfort, In The United Kingdom
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111145
Record Dates: First submitted 2010-08-26; First posted 2010-09-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2011-06

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Real world; observational; retrospective; database analysis
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Xalacom; Duotrav; Ganfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fixed dose prostaglandin combination
  Interventions: Drug: XALACOM; Drug: Duotrav; Drug: Ganfort

INTERVENTIONS:
Drug: XALACOM — Xalacom eye drops
Drug: Duotrav — Duotrav eye drops
Drug: Ganfort — Ganfort eye drops

SUMMARY:
The hypothesis is that there is no difference in persistency between Xalacom and the alternative fixed dose combination products (Duotrav and Ganfort) over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had received a prescription for either Xalacom, Ganfort and DuoTrav
* Greater than 18 years old
* Diagnosed with glaucoma or ocular hypertension
* Registered at the primary care practice for > 12 months

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had received a prescription for either Xalacom, Ganfort and DuoTrav, > 18 years old, diagnosed with glaucoma or ocular hypertension, registered at the primary care practice for > 12 months
Sampling Method: Non-Probability Sample
Enrollment: 2015 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Frequency distribution of persistent and non-persistent patients across study cohorts | 12 months
Frequency distribution of switchers, re-starters and discontinuing patients as well as patients commencing add-on therapy across the study cohorts | 12 months
Time to discontinuation of each cohort | 12 months

SECONDARY OUTCOMES:
Age and sex: Townsend Score of social deprivation, time since first THIN diagnosis of glaucoma or ocular hypertension | 12 months
Procedures: Laser, Trabeculectomy, viscocanalostomy, deep sclerectomy | 12 months
Ocular Pharmacological Treatments: Beta-blockers and Alpha-agonists | 12 months
Prostaglandin mono-therapies | 12 months
The cohort of patients which were evaluated in this study were investigated for the presence of history of disease for asthma, cardiovascular disease, diabetes, renal failure and systemic hypertension. The number of patients in each cohort were | 12 months
presented who had had (i) a 12 month history of any of the diseases or (ii) had had a history of any of the diseases. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111145&StudyName=Real%20World%20Data%20Study%20Assessing%20The%20Persistency%20Of%20Xalacom%20And%20The%20Other%20Fixed%20Dose%20Combination%20Products%2C%20Duotrav%20And%20Ganfort%2C%20In%20